CLINICAL TRIAL: NCT00127686
Title: Effect of Honey and Dextromethorphan on Nocturnal Cough and Sleep Quality for Coughing Children and Their Parents
Brief Title: Effect of Honey and Dextromethorphan on Nocturnal Cough and Sleep
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Honey Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 21163
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Cough; Respiratory Tract Infections
Keywords: cough; nocturnal cough; upper respiratory tract infection; sleep quality; childhood cough; Dextromethorphan; Honey
MeSH Terms: conditions — Cough; Respiratory Tract Infections; Sleep Initiation and Maintenance Disorders | interventions — Dextromethorphan

INTERVENTIONS:
Drug: Dextromethorphan
Drug: Buckwheat Honey

SUMMARY:
Cough is the most common reason for an acute care doctor's visit in the United States. Cough can affect sleep for both coughing children and their parents. The American Academy of Pediatrics does not endorse the use of dextromethorphan (DM), the most common over-the-counter (OTC) cough medication because of a lack of efficacy data and some potential for toxicity, particularly when taken in excess. In fact, DM has previously been shown to be no better than a placebo for cough in children. Therefore, alternative, therapeutic agents are needed. Honey anecdotally provides relief for symptoms due to upper respiratory tract infection (URI). This study seeks to use a survey to evaluate whether a single dose of honey and/or DM is better than no treatment at all for controlling nocturnal cough in children with URI and the effect of the treatments on sleep quality for coughing children and their parents. A single dose of honey or DM will be superior to no treatment for control of nocturnal cough due to upper URI as rated by both parents and children and will improve the sleep quality for those children and parents. Compared to DM, honey will be superior for controlling nocturnal cough due to upper URI (also based on child and parental report).

DETAILED DESCRIPTION:
Cough is one of the most common reasons for a doctor's visit in the United States and may be the most bothersome symptom for children with colds. It is particularly annoying at night because it can interrupt sleep for both coughing children and their parents. Dextromethorphan (DM), the most common over-the-counter (OTC) "cough medication," may not be as helpful for these symptoms as previously believed. Because of this, treatments are needed to better reduce the symptoms from a cold. Honey is a naturally occurring substance that may provide relief for cold symptoms. Children are being offered the opportunity to take part in this research because they have been diagnosed with a cold and have had difficulty sleeping due to their cough.

The purpose of this research is to use a survey to see if a single dose of honey or DM is better than no treatment at all for controlling nighttime cough in children, ages 2 to less than 18 years with a cold and if the medicine or honey helps the quality of sleep for the coughing children and their parents. DM has been approved by the Food and Drug Administration (FDA) and is available over the counter. The form of honey used in this study may also be purchased without a doctor's prescription.

About 125 male and female children from 2 to less than 18 years old will take part in this study at the Hershey Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 to <18 years
* Cough due to upper respiratory tract infection (URI), as determined by physical examination
* Sleep difficulty on the preceding night attributed to frequent cough
* Ability to swallow liquids
* Willingness of the child's guardian to participate in a survey

Exclusion Criteria:

* Signs/symptoms of more serious/treatable disease
* Itchy, watery eyes
* Frequent sneezing, tachypnea (respiratory rate >95th percentile) or labored breathing; symptoms for 8 or more days.
* History of asthma in the past 2 years
* Chronic lung disease, or seizure disorder
* Allergic reaction to honey or DM
* Selective serotonin reuptake inhibitors (SSRIs) or anti-malarial drugs
* Diabetes mellitus or signs/symptoms of insulin resistance

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2005-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Compared with no treatment, honey and DM will: improve the sleep quality for children with cough due to URI and improve the sleep quality for the parents of children with cough due to URI | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Paul, MD, MSc, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Paul IM, Beiler J, McMonagle A, Shaffer ML, Duda L, Berlin CM Jr. Effect of honey, dextromethorphan, and no treatment on nocturnal cough and sleep quality for coughing children and their parents. Arch Pediatr Adolesc Med. 2007 Dec;161(12):1140-6. doi: 10.1001/archpedi.161.12.1140. PMID 18056558
- See also: Pediatric Clinical Research Office: Penn State Milton S. Hershey Medical Center — http://www.hmc.psu.edu/pedsclinicalresearch/index.htm